CLINICAL TRIAL: NCT06519019
Title: Comparative Evaluation of Soft and Hard Tissue Healing and Implant Stability Of Hydrophilic Versus Conventional Titanium Dental Implants - A Randomized Clinical Trial.
Brief Title: Evaluation of Soft and Hard Tissue Healing and Implant Stability Of Hydrophilic Versus Conventional Titanium Dental Implants.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_147447
Record Dates: First submitted 2024-07-12; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Dental Implants
Keywords: Dental Implants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrophilic Dental Implant Group (Experimental): One dental implant placed will have hydrophilic properties.
  Interventions: Procedure: Dental Implant Surgery - Hydrophilic group
- Conventional Dental Implant Group (Active Comparator): This Conventional Dental implant group will act as control.
  Interventions: Procedure: Dental Implant Surgery - Conventional group

INTERVENTIONS:
Procedure: Dental Implant Surgery - Hydrophilic group — A full thickness mucoperiosteal flap was elevated, under Local anaesthesia, osteotomy sites were prepared according to manufactures instructions, and parallel pin was used to confirm position and angulation of osteotomy site. One site received a hydrophilic implant and the other site received a conventional implant.
  Ostell ISQ was used to measure primary stability of the dental implant. The surgical wound closure was with mattress and single interrupted sutures, using 4-0 vicryl suture.
  Arms: Hydrophilic Dental Implant Group
Procedure: Dental Implant Surgery - Conventional group — A full thickness mucoperiosteal flap was elevated, under Local anaesthesia, osteotomy sites were prepared according to manufactures instructions, and parallel pin was used to confirm position and angulation of osteotomy site. One site received a hydrophilic implant and the other site received a conventional implant.
  Ostell ISQ was used to measure primary stability of the dental implant. The surgical wound closure was with mattress and single interrupted sutures, using 4-0 vicryl suture.
  Arms: Conventional Dental Implant Group

SUMMARY:
Dental implants have become more common treatment for replacing missing teeth and aim to improve chewing efficiency, physical health and esthetic. Researchers always tried to improve design, mechanical and chemical properties of implant. Major benefit of surface modification are to improve hydrophilicity, cell to implant adhesion and cell proliferation. These modification improve osseointegration and reduce treatment duration. In this study investigators are evaluating healing capacity of hydrophilic implant compared to conventional implant.

DETAILED DESCRIPTION:
Implant stability at early stages is one of the most important factors affecting osseointegration success. Implant stability occurs as a result of mechanical engagement with the bone (primary stability), in addition to bone remodeling and regeneration (secondary stability) . Primary stability is certainly one of the fundamental criteria influencing implant success . Although there are several techniques to assess primary stability, one of the most popular digital methods is Resonance Frequency Analysis (RFA), Osstell® system (Osstell AB Stampgatan, Gotemborg, Sweden) and Periotest.® (Siemens Medical Systems Inc, Charlotte, Nc). The primary stability of implants also depends on the geometry of the implants (i.e., length, diameter, shape, and thread) besides the surgical technique, volume, and mechanical quality of local bone.

Several methods are widely used to modify the implant surface, such as sandblasting, acid etching, anodic oxidation, fluoride treatment, machining, titanium plasma spraying, and calcium phosphate coating. In dental implant, the surface treatment is used to modify the surface topography and surface energy, resulting in an improved wettability (hydrophilicity), increased cell proliferation and growth, and accelerated osseointegration process and reduced treatment duration. Hydrophilicity presents major advantages during the initial stages of wound healing and during the cascade of events that occurs during osseointegration, facilitating bone integration.

Although there are several studies which compares hydrophilic and hydrophobic implants, there are limited split mouth studies evaluating healing capacity of hydrophilic implants and hydrophobic implants.

Hence the aim of the present study is to evaluate the Marginal bone loss, healing of soft tissue, and primary and secondary implant stability of hydrophobic and hydrophilic implants in same subjects.

ELIGIBILITY:
Inclusion Criteria:

1. At least above 18 years of age.
2. Patients who needs replacement of two or more teeth in mandible.
3. Adequate bone volume to accommodate planned dental implants.

Exclusion Criteria:

1. General contraindication to dental implant treatment. (Uncontrolled diabetes and severe cardiovascular or infectious diseases).
2. Intravenous and oral bisphosphonate therapy.
3. Presence of severe, moderate or mild untreated periodontal disease.
4. Unwillingness to return for the follow-up examination.
5. Smokers.
6. Patients who are psychologically unable to participate.
7. Poor oral hygiene.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Implant Stability Using Resonance Frequency Analysis | "Baseline", "2 weeks", "1 month", "3 months"
  Implant stability is measured
Marginal Bone Loss Using RVG and Grid. | "3 months"
  Marginal Bone Loss Measured
Soft tissue healing | "1 Week", "2 weeks", "1 month", "3 months"
  Soft tissue healing will be assessed using Landry Turnbull and Howley Healing Index. Where soft tissue healing will be scored from 1 to 5, where score "1" indicate worse score and score "5" indicate Best score

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers.